CLINICAL TRIAL: NCT02821780
Title: CADASIL Disease Discovery
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160132; 16-H-0132
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-09-19

CONDITIONS: Germline Mutation in the NOTCH 3 Gene; Cardiovascular Disease; Arterial Stiffness; Pathogenesis of CADASIL; Clinical Phenotype of CADASIL
Keywords: Stroke; progressive white matter degeneration, and debilitating dementia.; progressive chronic hypoperfusion; Biospecimen Procurement; Laboratory Research Specimens; Natural History
MeSH Terms: conditions — Cardiovascular Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral autosomal dominant arteriopathy with subcortical infarct (CADASIL) is a lethal disease caused by a gene mutation that affects arteries in the brain. Symptoms include migraines, strokes, memory loss, and dementia. There are no treatments. Researchers want to study people who have CADASIL to learn more about it.

Objectives:

To learn more about CADASIL by studying people who have it.

Eligibility:

People ages 18-100 who were diagnosed with CADASIL in the past 5 years and can make their own decisions

Design:

Participants will be screened in another NIH protocol.

Participants will have 3 visits over 2 years. These may include:

* Physical exam
* Thinking and concentration tests
* Blood tests
* Skin biopsy: A small skin punch is removed from the arm or leg
* Eye exam and eye imaging tests
* Fluorescein angiogram: A catheter is placed in an arm vein. Dye is given through the catheter and travels

to the eyes.

* EndoPAT: A small clamp on the fingertip measures blood volume.
* Cardio-ankle vascular index (CAVI): Artery stiffness is tested with blood pressure cuffs on the arms and

legs. Soft electrodes on the skin measure heart signals.

* Brain MRI or MRA: They lie on a table that slides in and out of a tube that takes pictures. They may get

a contrast agent in their vein. It brightens the brain so researchers can see where blood flows.

* CT scan of the heart: They lie on a table that slides in and out of a machine that takes pictures.
* They get contrast dye injected through a catheter. They may get a medicine that makes their blood

vessels bigger or slows their heart rate.

DETAILED DESCRIPTION:
Small vessel diseases are conditions characterized by the narrowing of small arteries leading to an imbalance of blood supply upon demand. This results in a progressive chronic hypoperfusion with detrimental outcomes for the affected organ system and for the patient. Recent advances in genetic evaluation have identified several genetic variants causing cerebrovascular small vessel diseases. These diseases have common clinical presentation including recurrent strokes, progressive white matter degeneration, and debilitating dementia. The link between these pathologies is defects in the tunica media of arteries, which is composed mainly of vascular smooth muscle cells (vSMCs).

CADASIL (cerebral autosomal dominant arteriopathy with subcortical infarct and leukoencephalopathy) is caused by mutations in NOTCH3. The disease is of slow onset, with initial clinical manifestations in the third and fourth decade of life, but progressive and fatal. Predominant clinical features include migraine with aura (atypical or isolated), strokes, memory loss, and multiple psychiatric symptoms including dementia. Currently, CADASIL is considered the most common hereditary subcortical vascular dementia, however, treatments are palliative, and there is little prospect of future therapies to directly address causation and block progression. We propose to characterize the etiology and natural history of CADASIL subjects through comprehensive clinical and molecular characterizations. Subjects will be seen at the National Institutes of Health (NIH) once a year for a period of 2 years (total of 3 visits).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female, age 18 to 100 years (inclusive).
* Established diagnosis of CADASIL, as determined by genetic testing, in early stages of disease (0-5 years after diagnosis) with mild or no cognitive impairment.
* Willing and able to comply with study requirements.

EXCLUSION CRITERIA:

* Subjects unable to give informed consent without requirement for a legally authorized representative
* Subjects who decline to provide samples for blood and/or tissue studies, or who do not consent to have samples stored for future research
* Pregnant women are excluded due to study procedures (pregnancy test will be done in females of childbearing age under other NHLBI-approved protocols the subject is consented to, up to 48 hours prior to consenting to this protocol).
* Subjects unable to undergo an MRI scan

  * Subjects who have internal non-MRI compatible metals (i.e. cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or metal fragments in the eye) as these rendering an MRI unsafe
  * Subjects with ferromagnetic dental bridges or crowns (exclusion only for 7.0T)
  * Subjects unable to remain supine for the expected length of the MRI (i.e. up to 1 hour)
  * Subjects with uncontrolled head movements
  * Subjects who are claustrophobic for the expected length of the MRI (i.e. up to 1 hour) and claustrophobia cannot be controlled with anti-anxiety medication.
* Subjects whose scans or examinations show unexpected brain conditions.
* Subjects who do not speak English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, age 18 to 100 years (inclusive). Established diagnosis of CADASIL, as determined by genetic testing, in early stages of disease (0-5 years after diagnosis) with mild or no cognitive impairment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
To study the pathogenesis of CADASIL through comprehensive clinical evaluations and molecular studies on biospecimens collected under this protocol from affected and unaffected cohorts (as reference biospecimens). | 2 years
  pathogenesis of CADASIL through comprehensive clinical evaluations and molecular studies on biospecimens

SECONDARY OUTCOMES:
Clinical evaluations will be used to determine whether disease progression can be assessed. | 2 years
  Therefore, we will perform a comprehensive clinical and molecular assessment to determine possible correlations between clinical phenotypes, histological biopsy read-outs, and molecular findings

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Nationwide Children s Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0132.html